CLINICAL TRIAL: NCT04527055
Title: The Studies of Integrating Gastric and Gut Microbiota, F. Prausnitzii Metabolites, Microenvironment, and Epigenetics to Identify the Cancer Risk of H. Pylori-related Precancerous Conditions Through an AI System and Control the Risky by Probiotic Supplements
Brief Title: The Efficacy of 10-day and 14-day Bismuth-based Quadruple Therapy in First-line H. Pylori Eradication
Acronym: Bsm10
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Hsiu-Chi Cheng, Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-BR-109-012
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Helicobacter Pylori Infection; Dysbiosis; Probiotics
MeSH Terms: conditions — Dysbiosis | interventions — bismuth tripotassium dicitrate; Tablets; Lacteol; Esomeprazole; Metronidazole; Tetracycline

STUDY DESIGN:
Intervention Model Description: Among the H. pylori-infected patients, they are randomized to the 14-day bismuth-based quadruple therapy group and the 10-day bismuth-based quadruple therapy group to receive a 14-day and 10-day course, respectively, of the bismuth-based quadruple therapy. Afterward, the patients stop taking the proton pump inhibitor and antibiotics for 4 to 6 weeks, and then they receive 13C-UBT or an H. pylori stool antigen test to confirm successful eradication or not.
  Patients' fecal microbiota profiling is performed before and after H. pylori eradication. If patients have the depletion of gut F. prausnitzii 12 months after H. pylori eradication, they are enrolled to the probiotic supplement trial. They are randomized to the probiotic therapy group ingesting probiotic powder twice daily for 24 weeks and the non-probiotic control group, respectively.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- The 14-day bismuth-based quadruple therapy group (Active Comparator): The patients receive a 14-day course of the bismuth-based quadruple therapy, including esomeprazole (Nexium 40 mg) 1 tab twice a day, bismuth subcitrate (dibismuth trioxide) (KCB F.C. 120 mg) 1 tab four times a day, metronidazole (Flagyl 250 mg) 2 tab thrice a day, and tetracycline (250 mg) 2 tab four times a day.
  Interventions: Drug: Bismuth Subcitrate 120 MG Oral Tablet; Drug: Esomeprazole 40mg; Drug: Metronidazole 250 MG; Drug: Tetracycline Pill
- The 10-day bismuth-based quadruple therapy group (Active Comparator): The patients receive a 10-day course of the bismuth-based quadruple therapy, including esomeprazole (Nexium 40 mg) 1 tab twice a day, bismuth subcitrate (dibismuth trioxide) (KCB F.C. 120 mg) 1 tab four times a day, metronidazole (Flagyl 250 mg) 2 tab thrice a day, and tetracycline (250 mg) 2 tab four times a day.
  Interventions: Drug: Bismuth Subcitrate 120 MG Oral Tablet; Drug: Esomeprazole 40mg; Drug: Metronidazole 250 MG; Drug: Tetracycline Pill
- The non-H. pylori-infected control (No Intervention): Age- and sex-matched patients who do not have H. pylori infection by endoscopic gastric biopsy are enrolled as the non-H. pylori-infected control.
- The probiotic therapy group (Active Comparator): The patients who still have depletion of gut F. prausnitzii 12 months after H. pylori eradication are enrolled into the probiotic supplement trial. They are randomized to the probiotic therapy group ingesting probiotic powder twice daily for 24 weeks. The probiotic powder is named as "President AB powder", which contains an approximately equal mixture of Lactobacillus acidophilus and Bifidobacterium lactis Bb12 at a concentration of >= 10E9 CFU/mL (President Corp., Tainan, Taiwan).
  Interventions: Dietary Supplement: Lactobacillus acidophilus and Bifidobacterium lactis Bb12
- The non-probiotic control group (No Intervention): The patients who still have depletion of gut F. prausnitzii 12 months after H. pylori eradication are enrolled into the probiotic supplement trial. They are randomized to the non-probiotic control therapy and they do not ingest probiotic powder.

INTERVENTIONS:
Drug: Bismuth Subcitrate 120 MG Oral Tablet — Bismuth Subcitrate (120 MG Oral Tablet) 1 tab per oral four times per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: KCB F.C.
  Arms: The 10-day bismuth-based quadruple therapy group; The 14-day bismuth-based quadruple therapy group
Dietary Supplement: Lactobacillus acidophilus and Bifidobacterium lactis Bb12 — The probiotic powder per oral twice daily for 24 weeks. The probiotic powder is named as "President AB powder", which contains an approximately equal mixture of Lactobacillus acidophilus and Bifidobacterium lactis Bb12 at a concentration of >= 10E9 CFU/mL (President Corp., Tainan, Taiwan).
  Other Names: President AB powder
  Arms: The probiotic therapy group
Drug: Esomeprazole 40mg — Esomeprazole (40 mg) 1 tab per oral twice per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: Nexium
  Arms: The 10-day bismuth-based quadruple therapy group; The 14-day bismuth-based quadruple therapy group
Drug: Metronidazole 250 MG — Metronidazole (250 MG) 2 tab per oral thrice per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: Tolizole
  Arms: The 10-day bismuth-based quadruple therapy group; The 14-day bismuth-based quadruple therapy group
Drug: Tetracycline Pill — Tetracycline (250 MG) 2 tab per oral four times per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: Tetracycline (250 mg)
  Arms: The 10-day bismuth-based quadruple therapy group; The 14-day bismuth-based quadruple therapy group

SUMMARY:
Helicobacter pylori (H. pylori) infection is the major cause of gastritis, peptic ulcer disease, and gastric cancer in adults. Bismuth-based quadruple therapy is recommended by a recent review to be the first-line treatment for H. pylori eradication, replacing clarithromycin-based triple therapy. It is because the eradication rates of triple therapy in adults have declined due to increasing clarithromycin resistance. The best regimen for H. pylori eradication should be the one which succeeds on the first attempt. However, the effectiveness and the optimal duration of bismuth-based quadruple therapy for first-line H. pylori eradication in adults are unknown. Moreover, the impacts on gut microbiota after H. pylori eradication should be concerned; for example, bismuth-based quadruple therapy decreases F. prausnitzii richness. The transient perturbation of the gut microbiota after H. pylori eradication were restored at 8 weeks and one year in subjects receiving clarithromycin-based triple therapy but not fully recovered in those receiving bismuth-based quadruple therapy. Therefore, the important issues are that the short-term and long-term gut dysbiosis and the recovery of gut F. prausnitzii depletion in H. pylori-infected adult patients after bismuth-based quadruple therapy. It is also uncertain the role of irreversible gut dysbiosis even though H. pylori is eradicated in gastric persist inflammation and progress to cancer, and whether probiotics could be helpful in recovering gut dysbiosis.

The therapeutic strategy to eradicate H. pylori infection is based on antibiotics; however, this strategy not only increases drug resistant rates of the pathogen but also shapes the gut microbiota.

The investigators hypothesize that bismuth-based quadruple therapy could be an optimal regimen for first-line H. pylori eradication in the era of increasing clarithromycin resistance; moreover, gut dysbiosis could be reversed after bismuth-based quadruple therapy. Furthermore, the efficacy of the10-day course is not inferior to that of the 14-day course in H. pylori eradication. The investigators also hypothesize that probiotics could restore gastric or gut dysbiosis, especially gut F. prausnitzii depletion.

DETAILED DESCRIPTION:
Bismuth-based quadruple therapy is recommended by a recent review to be the first-line treatment for H. pylori eradication, replacing clarithromycin-based triple therapy. It is because the eradication rates of triple therapy in adults and clarithromycin-contained sequential therapy in children have declined due to increasing clarithromycin resistance in both adults and children. The best regimen for H. pylori eradication should be the one which succeeds on the first attempt. However, the effectiveness and the optimal duration of bismuth-based quadruple therapy for first-line H. pylori eradication in children and adults, respectively, are unknown. Moreover, the impacts on gut microbiota after H. pylori eradication should be concerned; nevertheless, the results are controversial.

Probiotic supplements are beneficial to gut health through modulation of the gut microbiota and metabolomics. Our previous studies also reported that the efficacy of H. pylori eradication is improved and relevant immune response could be modified by probiotics-containing yogurt ingestion. Our preliminary data have shown that gut F. prausnitzii depletion in H. pylori-infected children could be reversed after triple eradication therapy with probiotics-containing yogurt ingestion. However, it is uncertain whether the recovery of gut F. prausnitzii by probiotics could restore gut dysbiosis or improve systemic inflammation, and the role of gut F. prausnitzii or metabolites in the H. pylori-microbiota-host metabolism axis.

The investigators hypothesize that bismuth-based quadruple therapy could be an optimal regimen for first-line H. pylori eradication in the era of increasing clarithromycin resistance; moreover, gut dysbiosis could be reversed after bismuth-based quadruple therapy. Furthermore, the efficacy of the10-day course is not inferior to that of the 14-day course in H. pylori eradication. Among the H. pylori-infected patients, they are randomized to the 14-day bismuth-based quadruple therapy group and the 10-day bismuth-based quadruple therapy group to receive a 14-day and 10-day course, respectively, of the bismuth-based quadruple therapy, including esomeprazole (Nexium 40 mg) 1 tab twice a day, dibismuth trioxide (KCB F.C. 120 mg) 1 tab four times a day, metronidazole (Flagyl 250 mg) 2 tab thrice a day, and tetracycline (250 mg) 2 tab four times a day.

Moreover, the investigators also hypothesize that probiotics could restore gastric or gut dysbiosis, especially gut F. prausnitzii depletion. The patients who still have depletion of gut F. prausnitzii 12 months after H. pylori eradication are enrolled into the probiotic supplement trial. They are randomized to the probiotic therapy group ingesting probiotic powder twice daily for 24 weeks and the non-probiotic control group, respectively. The probiotic powder is named as "President AB powder", which contains an approximately equal mixture of Lactobacillus acidophilus and Bifidobacterium lactis Bb12 at a concentration of >= 10E9 CFU/mL (President Corp., Tainan, Taiwan)

Sample size assessment: The investigators propose that the eradication rates in the bismuth-based quadruple therapy are ~97%. The case ratio of the two groups is 1:1. If there is a true difference in favor of the 14-day bismuth-based quadruple therapy of 7% (10-day therapy vs. 14-day therapy, < 90% vs. 97%), then a total of 250 patients are required to be 90% (power) sure that the upper limit of a one-sided 97.5% confidence interval (or equivalently a 95% two-sided confidence interval) will exclude a difference in favor of the 14-day bismuth-based quadruple therapy group of more than 7% [Sealed Envelope Ltd. 2012. Power calculator for binary outcome non-inferiority trial. [Online] Available from: https://www.sealedenvelope.com/power/binary-noninferior/ [Accessed Sun Feb 14 2021]. Assuming a surveying failure rate of ~20%, at least 312 patients are needed.

In addition, the investigators propose that the rates of gut F. prausnitzii depletion before and after probiotic therapy are 50% and 25%, respectively. With a two-side alpha value of 0.05 and power of 80% (β=0.20), the number of patients required is 92 in such a paired sample. Assuming a surveying failure rate of 10%, at least 103 subjects are needed in the probiotic therapy group. Moreover, according to case ratio of the probiotic therapy group and the non-probiotic control group as 7:3, and the number required is 46 in the non-probiotic control group.

Statistical analysis: The statistical analysis is performed with SPSS software (SPSS 17, Chicago, IL, USA). The Student's t-test, Pearson's χ2 test, and Mann-Whitney U test are conducted to identify the statistical differences between the two comparison groups. One-way ANOVA with Tukey's least significant difference, Pearson's χ2 test, and Kruskal-Wallis one-way ANOVA by ranks and post hoc comparison by Mann-Whitney U test are used to identify the statistical differences between the three or more comparison groups. Paired t-test, McNemar, and Wilcoxon signed-rank test are conducted to identify the statistical differences between the pair data. All of the tests are two-tailed with the statistical significance defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are > 18 years
* Receive gastroscopy because of dyspepsia, acid regurgitation, melena, hematemesis, or others

Exclusion Criteria:

* Bleeding diathesis,
* Major organic diseases
* Malignancy
* Diseases treated with chemotherapy within one month
* Diseases treated with steroids within one month
* Diseases treated with antibiotics within one month,
* Users of aspirin within four weeks before enrollment
* Users of nonsteroidal anti-inflammatory drugs within four weeks before enrollment
* Users of cyclooxygenase-2 selective inhibitors within four weeks before enrollment
* History of H. pylori eradication
* Ingest probiotics or probiotics-containing yogurt with a frequency of >= twice per week one month prior to enrollment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The successful eradication rate | About 4 to 6 weeks after receiving the H. pylori eradication regimen
  The patients stop taking the proton pump inhibitor and antibiotics for 4 to 6 weeks, and then they receive 13C-UBT or an H. pylori stool antigen test to confirm successful eradication or not.

SECONDARY OUTCOMES:
Adverse effects and adherence to medications of the 10-day bismuth-based quadruple therapy and 14-day bismuth-based quadruple therapy groups | About 2 to 4 weeks after receiving the H. pylori eradication regimen
  Secondary endpoints are the rates of adverse events and medication adherence. Adverse events and medication adherence are assessed by physicians and format questionnaire survey after completing treatment. Good adherence to medications is defined of taking >= 80% of medications. Adverse events include dizziness, skin rash, headache, unpleasant taste, abdominal pain, nausea, vomiting, diarrhea, constipation, abdominal fullness, glossitis, darkened stool, fatigue, and anorexia. Adverse events are divided into mild (no daily activity restricted) and severe (daily activity restricted or unable to work).
Fecal microbiota and metabolites and the microbial evolution after H. pylori eradication | Baseline, 6-12 months after receiving the H. pylori eradication regimen or after endoscopy
  We enroll subjects who are H. pylori-infected and stages III-IV of either OLGA or OLGIM into the high-risk group; subjects who are H. pylori-infected, stages 0-II of both OLGA and OLGIM, and age- and sex-matched for the high-risk group into the low-risk group; and subjects who are H. pylori negative, stages 0-II of both OLGA and OLGIM, and age- and sex-matched for the high-risk group into the control group.
  Bacterial taxanomy and metabolites are analyzed by 16S full-length rRNA sequencing and UHPLC with electrospray ionization.
  We compare the differences of fecal microbiota between the H. pylori-infected and control groups.
  We identify microbes with abundance difference between the high-risk and control groups, between the low-risk and control groups, and between the high-risk and low-risk groups.
  We compare the evolutionary changes of fecal microbiota between baseline, 2, 6-12 months after H. pylori eradication. We explore the fecal microbiota which mediates metabolites.
Fecal inflammatory parameters and their evolution after H. pylori eradication | Baseline, 2, 6, 9, and 12 months after receiving the H. pylori eradication regimen or after endoscopy
  The supernatant of stool is tested by ELISA for sIgA, interleukin 6 (IL-6), IL-10, and TGF-β (Quantikine; R&D Systems, Minneapolis, MN). Fecal lactoferrin and calprotectin are measured using a commercial Leuko-Test kit (TechLab, Blacksburg, VA) and PhiCal Fecal Calprotectin Immunoassay kit (Genova Diagnostics, Asheville, NC), respectively.
Gastric microbiota and its evolution after H. pylori eradication | The patients receive surveillance endoscopy one year after H. pylori eradication
  Gastric fresh mucosa is biopsied for microbiota survey at surveillance endoscopy. The differences of gastric microbiota are compared at baseline and after H. pylori eradication in the H. pylori-infected group.
Gastric precancerous conditions and the evolution after H. pylori eradication | About 12 months after H. pylori eradication
  To validate the evolution of gastric precancerous conditions, patients are divided into six groups, including normal, CGI, SPEM, stages I-II of both Operative Link for Gastritis Assessment (OLGA) and Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM), advanced stages (III-IV) of either OLGA or OLGIM, and dysplasia according to the Correa's cascade. The study plans to compare the evolution of the steps of Correa's cascade after H. pylori eradication.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chi Cheng, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Helicobacter pylori study group, National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang EH, Chen WY, Chiang HC, Li CH, Wu IH, Chen PJ, Wu CT, Tsai YC, Cheng WC, Huang CJ, Sheu BS, Cheng HC. 10-Day versus 14-day bismuth quadruple therapy for first-line eradication of Helicobacter pylori infection: a randomised, open-label, non-inferiority trial. EClinicalMedicine. 2024 Mar 11;70:102529. doi: 10.1016/j.eclinm.2024.102529. eCollection 2024 Apr. PMID 38500841
- [Derived] Cheng HC, Yang YJ, Yang HB, Tsai YC, Chang WL, Wu CT, Kuo HY, Yu YT, Yang EH, Cheng WC, Chen WY, Sheu BS. Evolution of the Correa's cascade steps: A long-term endoscopic surveillance among non-ulcer dyspepsia and gastric ulcer after H. pylori eradication. J Formos Med Assoc. 2023 May;122(5):400-410. doi: 10.1016/j.jfma.2022.11.008. Epub 2022 Nov 30. PMID 36463082